CLINICAL TRIAL: NCT03678662
Title: The Influence of Expectations Induced by Information Prior to Exercise on the Change in Pain Perception After a 3 Min Wallsquat Exercise in Healthy Subjects: A Randomized Controlled Trial.
Brief Title: Influence of Expectations on Change in Pain Perception After a 3 Min Wallsquat Exercise.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Odense University Hospital (Other)
Collaborators: University of Southern Denmark (Other)
Responsible Party: Principal Investigator, Peter Thinggaard, Stud. M.Sc. Physiotherapy, Odense University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 62039
Record Dates: First submitted 2018-09-12; First posted 2018-09-19 (Actual); Last update posted 2018-11-26 (Actual); Status verified 2018-11

CONDITIONS: Pain; Physical Activity
Keywords: Exercise-induced hypoalgesia, expectation, pain sensitivity
MeSH Terms: conditions — Pain; Motor Activity

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Participants will not be aware of which group they are allocated to. The experimenter who is assessing pressure pain threshold and tolerance is blinded to the study group of the participant.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- hyperalgesia expectation (Experimental): In this group the subjects will be told that the 3 minutes wall squat will have pain-enhancing effects.
  Interventions: Other: Neutral
- hypoalgesia expectation (Experimental): In this group the subjects will be told that the 3 minutes wall squat will have pain-diminishing effects.
  Interventions: Other: Hypoalgesia expectation
- Neutral (Active Comparator): In this group the subjects expectations are not manipulated
  Interventions: Other: Hyperalgesia expectation

INTERVENTIONS:
Other: Hypoalgesia expectation — "Before and after the squat exercise, assessment of how you experience pressure pain with the 2 devices you have just become acquainted with will be repeated. While doing the squat exercise you will be asked to indicate pain in the thigh muscles.
  What we currently know about the effect of exercise on the experience of pressure pain is that after eg. cycling or walking, more pressure can be applied before the pressure starts to hurt and more pressure is required before you can't withstand anymore.
  Whether this applies to a squat exercise, as the one you are about to perform, has not yet been investigated, but we expect that the same applies here, namely, that more pressure is required before you feel the pressure begins to hurt you and you will be able to endure a greater pressure."
  Supported by visual information.
  Other Names: Randomization group a
  Arms: hypoalgesia expectation
Other: Hyperalgesia expectation — "Before and after the squat exercise, assessment of how you experience pressure pain with the 2 devices you have just become acquainted with will be repeated. While doing the squat exercise you will be asked to indicate pain in the thigh muscles.
  What we currently know is that exercise can cause muscle pain, both during and after training. You may have experienced muscle soreness yourself in relation to training? We expect that the same will apply here. Namely, after performing this squat exercise, which will likely hurt your thigh muscles while doing it, you will experience that the pressure applied afterwards, with the two devices you have just become acquainted with, should be less before it starts to hurt and that you can endure less pressure."
  Supported by visual information.
  Other Names: Randomization group b
  Arms: Neutral
Other: Neutral — "Soon you are going to do a training exercise in a squat position up against the wall for 3 min. Following the squat exercise, we will repeat the measurement of how you experience pressure pain with the 2 devices you have just become acquainted with. While doing the squat exercise you will be asked to indicate pain in the thigh muscles."
  Other Names: Randomization group c
  Arms: hyperalgesia expectation

SUMMARY:
The purpose of this study is to investigate how expectations induced by information given prior to exercise influence the magnitude of exercise-induced hypoalgesia after a 3 min wallsquat exercise in healthy subjects. The study is a double blinded (participant, investigator) randomized controlled trial The results from the study may be of great importance to the understanding of exercise-induced hypoalgesia, and whether the information related to exercise as pain relief can be used in practice for patients with pain.

The subjects are randomized to 1 in 3 groups. Hypoalgesia expectation, hyperalgesia expectation, neutral expectation. Each group (besides the neutral group) is given different information of what to expect on pain ratings after a 3 minutes wallsquat.

DETAILED DESCRIPTION:
Painful conditions are a major societal and economic problem and in Denmark, almost every fifth person suffers from long-lasting pain. Effective treatment of these conditions is vital not only to alleviate the pain but also to prevent repeated episodes of personal disorder and impaired work ability. Based on the hypothesis that physical activity and exercise lead to a change in pain perception, Pain Center South, Odense University Hospital has conducted a series of research projects which have investigated the immediate effect of various types of acute exercise on the pain sensitivity of both healthy subjects, patients with chronic pain in the knee and in patients with more 'complex' chronic pain who were referred to treatment at the Pain Center. The results showed that healthy subjects achieved a reduced overall pain sensitivity after both high intensity aerobic exercise (cycling) and low and high intensity isometric training (strength-like exercise on the arm and leg). This phenomenon is called 'exercise-induced hypoalgesia' or 'training-induced pain relief'. A recently published study from Australia has also shown that the effect of exercise can be positively influenced by the information given prior to exercise, indicating that some of the experience of exercise may be related to expectations of the effect. This may be one of the reasons why patients with chronic pain do not experience a positive effect, as opposed to healthy people, as chronic pain patients may previously have experienced no effect of exercise or perhaps even worsening / flareup in post-workout pain.

The purpose of this study is to investigate how expectations induced by information given prior to exercise influence the magnitude of exercise-induced hypoalgesia after a 3 min wallsquat exercise in healthy subjects. The pain sensitivity of the deep structures is investigated with two different pressure-gauges for the testing of mechanical pressure pain sensitivity. Pain sensitivity is examined on the leg and arm before and after the exercise. Pressure-sensitivity is evaluated using a handheld pressure-algometer for testing mechanical pressure pain-threshold in the deeper musculoskeletal structures. The pain-threshold is evaluated on the thigh and shoulder.

To investigate additional facets of pain-sensitivity, computer-controlled cuff geometry is used. The computer-controlled cuff algorithm is less affected by local differences in pain sensitivity to the handheld pressure algometer and the cuff algorithm can also affect a larger portion of the deep tissue than the pressure algometer can.

The cuff gauge consists of a blood pressure cuff placed around one lower leg and then slowly inflated. The pain response is registered continuously and the stimulus response function can then be established. The cuff algorithm has a maximum pressure that ensures no tissue damage to the subject and the device is automatically stopped at 100 kPa. Both the handheld pressure gauge and the cuff algorithm have proven to be a valid and reliable techniques for investigating the pain-sensitivity of healthy subjects.

The person performing the measurements before and after the exercise is blinded to what information the subject has received, likewise the patient is blinded to the group randomization.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects without current recurrent or prolonged painful diseases.
* The subjects should speak and understand Danish.

Exclusion criteria:

* Pregnancy
* Previous addictive behavior defined as abuse of hash, opioids or other euphoric substances.
* Previous painful or mental illnesses, neurological or circulatory diseases in the form of heart or lung disease.
* Lack of co-operation.
* Subjects who perform elite sports.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 83 (Actual)
Dates: Start 2018-09-19 (Actual); Primary Completion 2018-11-22 (Actual); Study Completion 2018-11-22 (Actual)

PRIMARY OUTCOMES:
Pressure pain threshold | At baseline before randomization and after the 3 minutes wallsquat - Day 1
  Between group comparison of the primary outcome, change in pressure pain threshold from baseline to post test. Pressure pain threshold is measured with a cuff algometer and pressure algometer respectively. Pressure pain threshold is measured in Kilopascal with rising pressure from 0 to infinity Kilopascal on the pressure algometer and from 0 to 100 Kilopascal on the cuff algometer. The cuff algometer is self-administered by the subject with a handheld joypad illustrating a Visual Analog Scala. Pressure pain threshold is registered in the computer when the subject reaches 0.1 centimeter and 1 centimeter on Visual Analog Scala on the joypad.
Pressure pain tolerance | At baseline before randomization and after the 3 minutes wallsquat - Day 1
  Between group comparison of the primary outcome, change in pressure pain tolerance from baseline to post test.. Pressure pain tolerance is measured with a cuff algometer. Pressure pain tolerance is measured in Kilopascal with rising pressure from 0 to 100 Kilopascal. The cuff algometer is self-administered by the subject with a handheld joypad illustrating a Visual Analog Scala. Pressure pain tolerance is registered in the computer when the subject reaches 10 centimeter on Visual Analog Scala on the joypad. If the 100 kilopascal on the cuff algometer is reached before the subjects maximum tolerance, the present score on Visual Analog Scala is assessed.

SECONDARY OUTCOMES:
Retrospective expectation for hypoalgesia and hyperalgesia after 3 minutes wall squat. | Post-test score at day 1 (immediately after the last pain rating)
  Three item self-reported questionaire about the subjects retrospective expectations to change in pain ratings for pain tolerance and for pain threshold at both sites (quadriceps and trapezius) after a 3 minutes wall squat. The questionaire is retrospective and will be used after all test procedures is done and therefore not indicate the subjects prospective expectation. The questions will be scored from -10 to +10. Whereas -10 indicates the subjects retrospective expectations of much more pain and +10 indicates the subjects retrospective expectations of much less pain.
Numeric Pain Rating Scale (NPRS) | Test score at day 1 (during the 3 minute wall squat)
  Between group comparison of maximum pain intensity. Pain intensity is measured on Numeric Pain Rating Scale (NPRS) during wall squat. The NPRS is a segmented numeric pain scale in which the subject selects a whole number from 0 to 10 that best reflects the intensity of his/her pain. Whereas 0 is no pain and 10 is the worst possible pain.
International Physical Activity Questionaires (IPAQ) | Pre test, baseline - day 1
  The IPAQ is suitable for adults between 15 and 69 years of age and is used for sample surveillance of physical activity levels.

CONTACTS AND LOCATIONS:
Overall Officials: Gitte Handberg, MD, Study Director — Pain Center, OUH
Locations (1):
- Pain Center South, Odense, Fyn, Denmark

REFERENCES:
- [Derived] Vaegter HB, Thinggaard P, Madsen CH, Hasenbring M, Thorlund JB. Power of Words: Influence of Preexercise Information on Hypoalgesia after Exercise-Randomized Controlled Trial. Med Sci Sports Exerc. 2020 Nov;52(11):2373-2379. doi: 10.1249/MSS.0000000000002396. PMID 32366799